CLINICAL TRIAL: NCT07386392
Title: Effect of Medical Hypnosis Compared to Virtual Reality or Standard Care on Anxiety During Induction Treatment for Acute Myeloid Leukemia
Brief Title: Effect of Hypnosis and Virtual Reality on Anxiety During Treatment for Acute Myeloid Leukemia
Acronym: HYPNO-RV LAM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Association Laurette Fugain (Unknown); Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/22/0010
Record Dates: First submitted 2026-01-26; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Virtual reality; Anxiety; Chemotherapy; Post-traumatic stress; Quality of life; Supportive care
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anxiety Disorders | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hypnose (Experimental): Patients participate in six hypnosis sessions, each lasting 30 minutes, twice during the first and second weeks, then once a week for the following two weeks
  Interventions: Other: Hypnosis
- Virtual Reality (Experimental): Patients participate in nine virtual reality sessions, each lasting 20 minutes, three times during the first week, then twice a week for the following three weeks
  Interventions: Other: Virtual Reality
- Control (No Intervention): Patients do not receive hypnosis sessions or virtual reality sessions

INTERVENTIONS:
Other: Hypnosis — Each session is based on the hypnosis techniques described by Erickson. In general, a session includes a hypnotic induction phase, a period of deepening and suggestions specific to the symptoms, followed by a return to reality. The hypnotherapist will be someone outside the team, trained in the Ericksonian method, who will intervene at a specific time during the sessions.
  Arms: Hypnose
Other: Virtual Reality — Each patient will be able to choose their environment from among those available (forest, beach, Zen garden, scuba diving, winter landscape, northern lights, astral travel, Antarctica, Maldives, desert), accompanied by ambient sounds. During the sessions, patients will be seated in their rooms at a quiet time outside of any treatment.
  Arms: Virtual Reality

SUMMARY:
This is a pilot study comparing 3 arms (standard care with hypnosis / standard care with virtual reality / standard care alone), aimed at measuring the effect on anxiety during the induction treatment. Acute myeloid leukemia is considered an oncological emergency that requires chemotherapy treatment with a high risk of serious adverse effects due to prolonged bone marrow failure or drug toxicity. This situation is very stressful for patients, who must cope with the initial symptoms, the diagnosis of a serious cancer, an urgent hospitalization (sometimes in intensive care) and prolonged hospitalization, invasive procedures for diagnosis and initiation of treatment, and intensive chemotherapy requiring protective isolation to contain the risk of life-threatening infection. Added to this care context is the breakdown of family ties as well as socio-professional ties, generating major anxiety and a risk of post-traumatic stress disorder (symptoms, which are common in acute myeloid leukemia. The hypothesis of our study is that hypnosis and virtual reality sessions combined with standard care could reduce anxiety and enhance chemotherapy treatment in acute myeloid leukemia patients when they first learn of their diagnosis.

DETAILED DESCRIPTION:
Patients will be randomly assigned to one of the three arms. All patients will receive standard conventional chemotherapy treatments in accordance with international recommendations and standard conventional care (including supportive care) during their hospital stay. Depending on the group to which they are assigned, they will also participate in hypnotherapy or virtual reality sessions during their hospital stay. Patients will be asked to complete various self-administered questionnaires to measure their levels of anxiety, quality of life, and stress during the course of treatment, according to the study schedule

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18
* Patient diagnosed with acute myeloid leukemia in Western Occitanie
* Eligible for first-line induction chemotherapy with anthracycline and cytarabine
* Patient able to understand and respond to a self-administered questionnaire
* Affiliated with or beneficiary of a social security system
* Having signed the research consent form

Exclusion Criteria:

* Patients diagnosed with acute myeloid leukemia 3
* Patients who were treated in intensive care prior to hospitalization for induction therapy or following induction therapy
* Patients with a diagnosed chronic pain-inducing disease (e.g., rheumatoid arthritis), if not stable
* Patients with a confirmed diagnosis of psychopathology such as psychosis, depression, or burnout, if not stable
* Patients suffering from epilepsy, whether treated or not, or with a history of epilepsy
* Patients under guardianship, conservatorship, or legal protection
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of an intervention combining standard care and virtual reality on the anxiety levels of patients at the end of induction chemotherapy for acute myeloid leukemia, compared to standard care and standard care with hypnosis | 35 days
  Change in anxiety score, measured using the Hospital Anxiety and Depression Scale

SECONDARY OUTCOMES:
Effect of an intervention combining standard care and virtual reality, compared to standard care and standard care with hypnosis, on nociceptive pain | 35 days
  Pain will be measured using a numerical pain scale at inclusion (first day of hospitalization)
Evaluate the effect of an intervention combining standard care and virtual reality, compared to standard care and standard care with hypnosis, on anxiety | 3 months
  Change in anxiety scores using the Hospital Anxiety and Depression Scale
Evaluate the effect of an intervention combining standard care and virtual reality, compared to standard care and standard care with hypnosis, on quality of life | 3 months
  Quality of life scores using the specific Fact-Leu questionnary
Evaluate the effect of an intervention combining standard care and virtual reality, compared to standard care and standard care with hypnosis, on post-traumatic stress disorder | 3 months
  Post-traumatic stress disorder using the Posttraumatic Stress Disorder Checklist Scale
Evaluate the effect of an intervention combining standard care and virtual reality, compared to standard care and standard care with hypnosis, on remission rate | 35 days
  Remission rate by sternal puncture, performed systematically (as part of routine care). A blast count of less than 5% will indicate remission
Evaluate the effect of an intervention combining standard care and virtual reality, compared to standard care and standard care with hypnosis, on minimal residual disease | 35 days
  Minimal Residual Disease, using molecular biology or flow cytometry
Evaluate the effect of an intervention combining standard care and virtual reality, compared to standard care and standard care with hypnosis, on consumption of analgesics and psychotropic drugs | 35 days
  Medication consumption based on cumulative doses and the number of days on analgesics and psychotropic drugs
Evaluate the effect of an intervention combining standard care and virtual reality, compared to standard care and standard care with hypnosis, on occurrence of adverse events related to induction treatment | 35 days
  Adverse events related to induction treatment of Common Terminology Criteria for Adverse Events grade ≥ 3, as well as adverse events related to induction treatment such as nausea, vomiting, mucositis, diarrhea, weight loss, and alopecia, regardless of grade

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne TAVITIAN, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- IUCT Oncopole, Toulouse, France, France